CLINICAL TRIAL: NCT01929148
Title: Is Prophylactic Bilateral Salpingectomy Added to Laparoscopic Myomectomy as New Preventive Strategy for Ovarian Cancer a Safe Procedure?
Brief Title: Prophylactic Bilateral Salpingectomy and Laparoscopic Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor, University Magna Graecia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBS_myomectomy
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Abnormal Uterine Bleeding, Unspecified
Keywords: risk-reducing salpingectomy; prophylactic bilateral salpingectomy; ovarian cancer prevention; ovarian reserve
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic myomectomy plus PBS (Experimental): A Laparoscopic myomectomy plus Prophylactic bilateral salpingectomy will be performed in women which have accomplished their reproductive desire
  Interventions: Procedure: Prophylactic bilateral salpingectomy
- Laparoscopic myomectomy without PBS (Active Comparator): A standard laparoscopic myomectomy without any prophylactic salpingectomy will be performed
  Interventions: Procedure: Laparoscopic myomectomy without PBS

INTERVENTIONS:
Procedure: Prophylactic bilateral salpingectomy — Salpingectomy will be performed by coagulation and section of the tube, beginning from the very distal fimbrial end, carefully preserving the ovarian vascularization, and proceeding toward the uterine cornu
  Other Names: PBS, bilateral salpingectomy
  Arms: Laparoscopic myomectomy plus PBS
Procedure: Laparoscopic myomectomy without PBS — Standard laparoscopic myomectomy without salpingectomy
  Other Names: LM
  Arms: Laparoscopic myomectomy without PBS

SUMMARY:
We already demonstrated that the addiction of PBS to Total Laparoscopic Hysterectomy (TLH) has no negative effects in term of ovarian function, evaluated by anti-Müllerian hormone (AMH), Follicle Stimulating Hormone (FSH), Antral Follicle Count (AFC), mean ovarian diameters and Peak Systolic Velocity (PSV). In addition, in our experience, no negative surgical outcomes (in terms of operative time, intraoperative blood loss, postoperative hospital stay, postoperative return to normal activity and complication rate) are related to PBS step in TLH.

Although the good statistical reliability of our retrospective data, we want to prospectively confirm our results. Moreover we aim to refine PBS safety demonstration by collecting also 3D ultrasound parameters [AFC, ovarian volume (OV), Vascularization Index (VI), Flow Index (FI) and Vascularization Flow Index (VFI)]. Hormonal and ultrasonographic parameters may possibly be unified into a new diagnostic algorithm (already at an advanced stage of production in UMG Department) able to estimate the ovarian function both in term of reproductive ability that in term of distance from menopause.

DETAILED DESCRIPTION:
We will enroll the first 77 patients who will agree to implement PBS to laparoscopic myomectomy (LM) (study group), starting from September 1, 2013. Other 77 patients who will ask us to undergo LM without the addiction of PBS will constitute the control group. For each patient, ovarian reserve modification before and after surgery will be recorded as the primary outcome. Specifically, one month before and three months after laparoscopy, on day 1 to 4 of menstrual cycles serum AMH, FSH and E2 will be evaluated and a transvaginal ultrasound examination (Voluson E8 Expert or Voluson-i - GE Healthcare Ultrasound) to assess AFC, OV, VI, FI and VFI, will be carried out by the same experienced ultrasonographist responsible for the ambulatory of ovarian reserve in each Unit.

Ovarian reserve modification will be defined as the difference (expressed as Δ) between post-operative and pre-operative values of AMH, FSH, AFC, OV, VI, FI and VFI. For each surgical procedure, moreover, operative time, variation of hemoglobin level, postoperative hospital stay, postoperative return to normal activity and complication rate will be recorded as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Indication to laparoscopic myomectomy
* Accomplished reproductive desire

Exclusion Criteria:

* Age older than 50 years
* family history of ovarian cancer, BRCA positive
* basal FSH value of >20 IU/mL and/or E2 levels >60 pg/mL
* presence of menopausal symptoms,irregular (cycle-to-cycle variation over 12 months >20 days orpresence of any breakthrough bleeding) menstrual cycles, hormonereplacement treatment and/or hormonal contraception for the last 3 months, history of previous uterine or ovarian surgeries, and imaging suggestive of ovarian cyst or tubal pathology at transvaginal ultrasound.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve modification | three months after laparoscopy
  Ovarian reserve modification will be defined as the difference (expressed as Δ) between post-operative and pre-operative values of anti-Müllerian hormone (AMH), Follicle Stimulating Hormone (FSH), Antral Follicle Count (AFC), Ovarian volume (OV), Vascularization Index (VI), Flow index (FI) and Vascularization Flow Index (VFI)

SECONDARY OUTCOMES:
Surgical outcomes | one day to one month after laparoscopy
  For each surgical procedure operative time, variation of hemoglobin level, postoperative hospital stay, postoperative return to normal activity and complication rate will be recorded as secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Md, PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Magna Graecia University - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro, CZ, Italy

REFERENCES:
- [Background] Morelli M, Venturella R, Mocciaro R, Di Cello A, Rania E, Lico D, D'Alessandro P, Zullo F. Prophylactic salpingectomy in premenopausal low-risk women for ovarian cancer: primum non nocere. Gynecol Oncol. 2013 Jun;129(3):448-51. doi: 10.1016/j.ygyno.2013.03.023. Epub 2013 Apr 2. PMID 23558052